CLINICAL TRIAL: NCT00347373
Title: Conjugated Linoleic Acid and Body Fat Mass in Obese Humans
Brief Title: Effect of Conjugated Linoleic Acid Supplement on Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: Cognis (Industry)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCRC2166
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Obesity
Keywords: conjugated linoleic acid; obesity; body composition; body fat mass; lean body mass
MeSH Terms: conditions — Obesity | interventions — Dietary Supplements

INTERVENTIONS:
Drug: Tonalin Conjugated linoleic acid (dietary supplement)

SUMMARY:
The purpose of this clinical trial is to examine the effects of a low and high dose of conjugated linoleic acid supplement on body composition in obese humans. Individuals with a body mass index between 30 and 35kg/m2 are randomized to receive either placebo, 3.2gCLA, or 6.4g CLA daily for twelve weeks. Changes in body composition, weight, and clinical laboratory values are compared between the three groups.

DETAILED DESCRIPTION:
Sixty healthy obese adult volunteers will be enrolled and randomized into either: 1) placebo, 2) 3.2 g CLA, or 3) 6.4 g CLA groups and supplemented for 12 weeks. Body fat mass (BFM) and lean body mass will be determined by DEXA at baseline and twelve weeks during the intervention. In addition, indirect calorimetry will be performed at baseline and twelve weeks to measure changes in energy expenditure. The effect of CLA supplementation on weight, waist and hip measurements, and BMI will also be determined at 12 weeks. Plasma CLA and pill counts will be measured as an indication of compliance. Several blood parameters will be monitored throughout the study, and five random 24-hour recall surveys will be used to monitor dietary intake of CLA-rich foods, energy, micronutrients and antioxidants.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 35 kg/m2

Exclusion Criteria:

* history of chronic disease
* food allergies or intolerances
* drug therapy for diagnosed disease or lipid-lowering
* use of weight-lowering medication or diet
* use of tobacco products
* current or planned pregnancy
* use of CLA supplement in previous 3 months
* current substance abuse
* abnormal clinical laboratory values

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2005-09

PRIMARY OUTCOMES:
Change in body fat mass at 12 weeks
Change in lean body mass at 12 weeks
Change in body mass index at 12 weeks
Change in body weight at 12 weeks
Change in energy expenditure at 12 weeks

SECONDARY OUTCOMES:
Change in lipid profile at 6 weeks and 12 weeks
Change in clinical laboratory values at 6 weeks and 12 weeks (safety)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Steck, PhD, MPH, RD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States